CLINICAL TRIAL: NCT06263244
Title: Specifying the Anti-inflammatory Effects of Ziltivekimab With Diverse Imaging Modalities and In-depth Cellular Phenotyping
Brief Title: Specifying the Anti-inflammatory Effects of Ziltivekimab
Acronym: SPIDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Prof. dr. E.S.G. Stroes, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL83403.018.22
Record Dates: First submitted 2023-08-03; First posted 2024-02-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Atherosclerosis; Inflammation
Keywords: DOTATATE; Ziltivekimab; Inflammation; Monocytes; CCTA; PET/CT
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — ziltivekimab

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After informed consent has been obtained, patients will be randomized via computer randomization to either 15 mg ziltivekimab (n=20) or placebo (n=20). On the eCRFs or other documents subjects will be identified by subject ID and randomization number only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ziltivekimab (Experimental): 15 mg ziltivekimab subcutaneously once per month for 5 months
  Interventions: Drug: Ziltivekimab
- Placebo (Placebo Comparator): Placebo, subcutaneously, once per month for 5 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Monoclonal antibody targeting IL-6
  Other Names: no other intervention name
  Arms: Ziltivekimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this randomized, double blind, placebo controlled trial is to study whether ziltivekimab therapy reduces arterial wall inflammation as assessed by imaging, and reduces the systemic inflammatory tone as assessed by circulating monocytes, inflammatory biomarkers and proteomics.

DETAILED DESCRIPTION:
Considering that ziltivekimab is currently undergoing a phase 3 CVOT trial, it is of great importance to elucidate its mechanistic effects. The objective of this study is to research whether ziltivekimab therapy for 20 weeks reduces arterial wall inflammation, as assessed by state-of-the-art imaging modalities, and reduces systemic inflammatory tone, as assessed by in depth phenotyping of circulating monocytes, inflammatory biomarkers and proteomics. The imaging modalities used in this study are 68Ga-DOTATATE PET/CT and CCTA. This study is designed as a single center, randomized, double-blinded, placebo-controlled intervention study in 40 atherosclerotic patients of 50 years and older with hsCRP levels of 2 mg/L and above.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older.
* Multi-vessel coronary artery disease (defined as CAD-RADS ≥2).
* Serum hsCRP level ≥2 mg/L.

Exclusion Criteria:

* Coronary stents in situ.
* Chronic or recent (<1 month) (serious) infections and/or clinical signs of acute (serious) infection.
* History of severe auto-immune diseases, or other (severe) (recurrent or chronic) inflammatory disorders.
* Use of preventive systemic antibiotics (antibiotics used to treat latent tuberculosis are exempted).
* Stable lipid lowering treatment for less than 4 weeks, including statins, ezetimibe and PCSK9 inhibition.
* Untreated latent tuberculosis, active hepatitis B (positive HBsAg and/or positive anti-HBc with detectable HBV DNA) or C, human immunodeficiency virus (HIV) not on stable antiretroviral regimen
* Uncontrolled diabetes (HbA1c >90 mmol/mol).
* Renal insufficiency, defined as eGFR <45 ml/min/1.73 m2.
* Platelet count <120,000 and >450,000 /mm3.
* Elevated liver enzymes (>3 ULN of liver transaminases), acute liver failure or known (severe) liver disease.
* Premenopausal women not using birth-control.
* History of gastrointestinal perforation, active diverticulitis (within 5 years) or active inflammatory bowel disease (within 12 months).
* Uncontrolled hypertension (systolic >180 mmHg; diastolic >110 mmHg).
* Diagnosis of (active) malignancy in last 5 years.
* Standard contra-indications to 68Ga-DOTATATE PET, and CT based on physician's experience and current practices.
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
TBRmax coronary arteries | 5.5 months
  mean percentage change in coronary arteries target to background ratio (TBRmax)
monocyte activation marker protein expression | 5.5 months
  The impact of ziltivekimab on a mass cytometry monocyte phenotype panel; expression markers such as CD14 and CD16.

SECONDARY OUTCOMES:
delta PCAT | 5.5 months
  Difference in PCAT (CCTA derived) after ziltivekimab treatment.
Correlation delta TBRmax and CCTA derived plaque characteristics | 5.5 months
  Correlation between changes in coronary 68Ga-DOTATATE uptake and anatomical plaque changes on CCTA.
delta SUVmax bone marrow | 5.5 months
  Difference in 68Ga-DOTATATE SUVmax of bone marrow after treatment.
delta TBRmax ascending aorta | 5.5 months
  Difference in 68Ga-DOTATATE TBRmax of ascending aorta after treatment
changes monocyte phenotype | 5.5 months
  The impact of ziltivekimab on monocyte phenotype in transendothelial migration (TEM) capacity and transcriptome profile.
changes in hsCRP | 5.5 months
  hsCRP (high-sensitivity C-reactive protein): mg/L
changes plasma cytokine and chemokine levels (pg/mL) | 5.5 months
  TNF-α (Tumor Necrosis Factor alpha): pg/mL IL-8 (Interleukin-8): pg/mL MCP-1 (Monocyte Chemoattractant Protein-1): pg/mL
changes plasma cytokine and chemokine levels (ng/mL) | 5.5 months
  sICAM (soluble Intercellular Adhesion Molecule): ng/mL sVCAM (soluble Vascular Cell Adhesion Molecule): ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: E.S.G. Stroes, Prof.dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No